CLINICAL TRIAL: NCT05606198
Title: Post-COVID-19 Monitoring in Routine Health Insurance Data With Focus on Autoimmune Diseases (POINTED-AD)
Acronym: POINTED-AD
Status: Completed | Type: Observational
Sponsor: Technische Universität Dresden (Other)
Collaborators: InGef - Institut für angewandte Gesundheitsforschung Berlin GmbH (Unknown); BARMER Institut für Gesundheitssystemforschung (bifg) (Unknown); Techniker Krankenkasse (Other); DAK Gesundheit (Other); AOK PLUS (Industry); IKK Classic (Unknown)
Responsible Party: Principal Investigator, Falko Tesch, Principal Investigator, Technische Universität Dresden
Other Study IDs: POINTED-AD
Record Dates: First submitted 2022-11-02; First posted 2022-11-04 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-07

CONDITIONS: Virus Diseases
MeSH Terms: conditions — Virus Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- COVID: 641,407 patients with a SARS-CoV-2 infection in the year 2020.
  Interventions: Other: Exposed to a SARS-CoV-2 infection
- Non-COVID: Matched patients with no SARS-CoV-2 infection during the study period.

INTERVENTIONS:
Other: Exposed to a SARS-CoV-2 infection — The study compared humans exposed to the SARS-CoV-2 infection with a matched group of those not exposed. No Intervention was applied.
  Groups: COVID

SUMMARY:
The SARS-CoV-2 (Severe acute respiratory syndrome coronavirus type 2) infection was in 2020 responsible for new disease related chronic conditions which have been referred to as Post-COVID. To date it is still unknown how common this condition is and how it might effect the working of the Immune system. The aim of the study is therefore to monitor the onset of autoimmune diseases in a large observational study consisting of German health insurance data.

DETAILED DESCRIPTION:
SARS-CoV-2 is a virus of the coronavirus family, which includes a large number of viruses that can cause a wide variety of diseases in humans. The SARS-CoV-2 virus causes acute symptoms associated with the infection and can cause chronic conditions known as Post-COVID. To understand how the virus might effect the working of the Immune system a large observational study of health insurance data from Germany was set up. The exposed patients were identified by a diagnosis indicating a confirmed laboratory test for COVID-19.

The basic question concerns the burden of the Post-COVID condition. The study investigate which autoimmune diseases or groups of autoimmune diseases are more common in humans after the exposure to the virus compared to a matched unexposed cohort. Further will this be investigated in subgroups of the population.

ELIGIBILITY:
Inclusion Criteria:

* At least one outpatient or inpatient diagnosis of COVID-19 with laboratory detection of the virus (ICD-10: U07.1!) in the year 2020
* Continuously insured with the respective health insurance between 2019-01-01/birth and 2021-06-30/death

Exclusion Criteria:

* Only an outpatient or inpatient diagnosis of COVID-19 without laboratory detection of the virus( ICD-10:U07.2!) till 30th of June 2021
* At least one outpatient or inpatient diagnosis of COVID-19 with laboratory detection of the virus (ICD-10: U07.1!) in the first half of the year 2021

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients were collected from six different health insurances/research institutions in Germany in the year 2020.
Sampling Method: Non-Probability Sample
Enrollment: 641407 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-25 (Actual); Study Completion 2023-06-19 (Actual)

PRIMARY OUTCOMES:
Incidence of Addison's disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Addison's disease recorded in outpatient or inpatient setting
Incidence of Alopecia areata | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Alopecia areata recorded in outpatient or inpatient setting
Incidence of Autoimmune hemolytic anemia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Autoimmune hemolytic anemia recorded in outpatient or inpatient setting
Incidence of Arteriitis temporalis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Arteriitis temporalis recorded in outpatient or inpatient setting
Incidence of Graves' disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Graves' disease recorded in outpatient or inpatient setting
Incidence of ankylosing spondylitis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of ankylosing spondylitis recorded in outpatient or inpatient setting
Incidence of Behcet's disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Behcet's disease recorded in outpatient or inpatient setting
Incidence of Churg-Strauss disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Churg-Strauss disease recorded in outpatient or inpatient setting
Incidence of Morbus Crohn | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Morbus Crohn recorded in outpatient or inpatient setting
Incidence of Dermatomyositis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Dermatomyositis recorded in outpatient or inpatient setting
Incidence of Diabetes type I | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Diabetes type I recorded in outpatient or inpatient setting
Incidence of Dermatitis herpetiformis (Duhring's disease) | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Dermatitis herpetiformis (Duhring's disease) recorded in outpatient or inpatient setting
Incidence of atopic dermatitis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of atopic dermatitis recorded in outpatient or inpatient setting
Incidence of Guillain-Barré-syndrome | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Guillain-Barré-syndrome recorded in inpatient setting
Incidence of Goodpasture syndrome | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Goodpasture syndrome recorded in outpatient or inpatient setting
Incidence of Hashimoto's thyroiditis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Hashimoto's thyroiditis recorded in outpatient or inpatient setting
Incidence of Autoimmune Hepatitis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Autoimmune Hepatitis recorded in outpatient or inpatient setting
Incidence of Juvenile rheumatoid arthritis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Juvenile rheumatoid arthritis recorded in outpatient or inpatient setting
Incidence of Kawasaki syndrome | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Kawasaki syndrome recorded in outpatient or inpatient setting
Incidence of Cutaneous lupus erythematosus | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Cutaneous lupus erythematosus recorded in outpatient or inpatient setting
Incidence of Cryoglobulinemia | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Cryoglobulinemia recorded in outpatient or inpatient setting
Incidence of Systemic lupus erythematosus | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Systemic lupus erythematosus recorded in outpatient or inpatient setting
Incidence of Morphea | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Morphea recorded in outpatient or inpatient setting
Incidence of Multiple sclerosis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Multiple sclerosis recorded in outpatient or inpatient setting
Incidence of Myasthenia gravis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Myasthenia gravis recorded in outpatient or inpatient setting
Incidence of Necrotizing vasculopathy | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Necrotizing vasculopathy recorded in outpatient or inpatient setting
Incidence of Bullous pemphigoid | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Bullous pemphigoid recorded in outpatient or inpatient setting
Incidence of Pemphigus vulgaris | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Pemphigus vulgaris recorded in outpatient or inpatient setting
Incidence of Polyarteritis nodosa | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Polyarteritis nodosa recorded in outpatient or inpatient setting
Incidence of Polymyalgia rheumatica | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Polymyalgia rheumatica recorded in outpatient or inpatient setting
Incidence of Polymyositis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Polymyositis recorded in outpatient or inpatient setting
Incidence of Psoriasis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Psoriasis recorded in outpatient or inpatient setting
Incidence of Idiopathic thrombocytopenic purpura | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Idiopathic thrombocytopenic purpura recorded in outpatient or inpatient setting
Incidence of rheumatoid arthritis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of rheumatoid arthritis recorded in outpatient or inpatient setting
Incidence of Sarcoidosis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Sarcoidosis recorded in outpatient or inpatient setting
Incidence of Sjögren's syndrome | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Sjögren's syndrome recorded in outpatient or inpatient setting
Incidence of Takayasu arteritis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Takayasu arteritis recorded in outpatient or inpatient setting
Incidence of Ulcerative colitis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Ulcerative colitis recorded in outpatient or inpatient setting
Incidence of Vitiligo | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Vitiligo recorded in outpatient or inpatient setting
Incidence of Wegener's disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of Wegener's disease recorded in outpatient or inpatient setting
Incidence of primary biliary cholangitis | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of primary biliary cholangitis recorded in outpatient or inpatient setting
Incidence of celiac disease | At least 12 weeks after the infection by SARS-CoV-2
  Incidence of a diagnosis of celiac disease recorded in outpatient or inpatient setting

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Schmitt, MD, MPH, Study Director — Center for Evidence-Based Healthcare, Technische Universität Dresden
Locations (1):
- Center for Evidence-Based Healthcare, Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tesch F, Ehm F, Vivirito A, Wende D, Batram M, Loser F, Menzer S, Jacob J, Roessler M, Seifert M, Kind B, Konig C, Schulte C, Buschmann T, Hertle D, Ballesteros P, Bassler S, Bertele B, Bitterer T, Riederer C, Sobik F, Reitzle L, Scheidt-Nave C, Schmitt J. Incident autoimmune diseases in association with SARS-CoV-2 infection: a matched cohort study. Clin Rheumatol. 2023 Oct;42(10):2905-2914. doi: 10.1007/s10067-023-06670-0. Epub 2023 Jun 19. PMID 37335408